CLINICAL TRIAL: NCT00344513
Title: Organized Program to Initiate Lifesaving Treatment in Hospitalized Patients With Heart Failure (OPTIMIZE-HF): An Internet-based Registry and Process of Care Improvement Program for Heart Failure Patients
Brief Title: Organized Program To Initiate Lifesaving Treatment In Hospitalized Patients With Heart Failure (OPTIMIZE-HF)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 105517/358
Record Dates: First submitted 2006-06-23; First posted 2006-06-26 (Estimated); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Heart Failure, Congestive
Keywords: registry; OPTIMIZE; Heart failure; OPTIMIZE-HF
MeSH Terms: conditions — Heart Failure | interventions — Angiotensin-Converting Enzyme Inhibitors

INTERVENTIONS:
Drug: Beta-blockers including Carvedilol
Drug: ACE inhibitors
  Other Names: Beta-blockers including Carvedilol

SUMMARY:
This program is designed to improve medical care and education of hospitalized patients with heart failure and accelerate the initiation of evidence-based heart failure guideline recommended therapies by administering them before hospital discharge. A registry component focusing on admission to discharge and 60- to 90-day follow-up is designed to evaluate the demographic, pathophysiologic, clinical, treatment, and outcome characteristics of patients hospitalized with heart failure.

ELIGIBILITY:
Inclusion criteria:

* Hospitalized for episode of worsening heart failure as primary cause of admission or significant heart failure symptoms that develop during the hospitalization when the initial reason for admission was not heart failure.
* Systolic dysfunction (LVEF < 40%) or heart failure symptoms in the setting of preserved systolic function (diastolic dysfunction).

Exclusion criteria:

* This study has no exclusion criteria.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50000
Dates: Start 2002-12-16 (Actual); Study Completion 2005-06-30 (Actual)

PRIMARY OUTCOMES:
Evaluate the number and percentage of eligible patients who are discharged on optimal therapy. Evaluate all HF indicators recommended by JCAHO and CMS.

SECONDARY OUTCOMES:
Mortality Recurrent hospitalization Number of patients receiving beta-blockers therapy within 60 to 90 days of initiation and mean beta-blocker dose 60-90 days following discharge.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

REFERENCES:
- [Derived] Patel K, Fonarow GC, Ekundayo OJ, Aban IB, Kilgore ML, Love TE, Kitzman DW, Gheorghiade M, Allman RM, Ahmed A. Beta-blockers in older patients with heart failure and preserved ejection fraction: class, dosage, and outcomes. Int J Cardiol. 2014 May 15;173(3):393-401. doi: 10.1016/j.ijcard.2014.03.005. Epub 2014 Mar 11. PMID 24703206
- [Derived] Mentz RJ, Wojdyla D, Fiuzat M, Chiswell K, Fonarow GC, O'Connor CM. Association of beta-blocker use and selectivity with outcomes in patients with heart failure and chronic obstructive pulmonary disease (from OPTIMIZE-HF). Am J Cardiol. 2013 Feb 15;111(4):582-7. doi: 10.1016/j.amjcard.2012.10.041. Epub 2012 Nov 29. PMID 23200803
- [Derived] Patel UD, Greiner MA, Fonarow GC, Phatak H, Hernandez AF, Curtis LH. Associations between worsening renal function and 30-day outcomes among Medicare beneficiaries hospitalized with heart failure. Am Heart J. 2010 Jul;160(1):132-138.e1. doi: 10.1016/j.ahj.2010.03.033. PMID 20598983
- [Derived] Hernandez AF, Greiner MA, Fonarow GC, Hammill BG, Heidenreich PA, Yancy CW, Peterson ED, Curtis LH. Relationship between early physician follow-up and 30-day readmission among Medicare beneficiaries hospitalized for heart failure. JAMA. 2010 May 5;303(17):1716-22. doi: 10.1001/jama.2010.533. PMID 20442387
- [Derived] Hernandez AF, Hammill BG, Peterson ED, Yancy CW, Schulman KA, Curtis LH, Fonarow GC. Relationships between emerging measures of heart failure processes of care and clinical outcomes. Am Heart J. 2010 Mar;159(3):406-13. doi: 10.1016/j.ahj.2009.12.024. PMID 20211302
- [Derived] Levy PD, Nandyal D, Welch RD, Sun JL, Pieper K, Ghali JK, Fonarow GC, Gheorghiade M, O'Connor CM. Does aspirin use adversely influence intermediate-term postdischarge outcomes for hospitalized patients who are treated with angiotensin-converting enzyme inhibitors or angiotensin receptor blockers? Findings from Organized Program to Facilitate Life-Saving Treatment in Hospitalized Patients with Heart Failure (OPTIMIZE-HF). Am Heart J. 2010 Feb;159(2):222-230.e2. doi: 10.1016/j.ahj.2009.11.009. PMID 20152220
- [Derived] Hernandez AF, Fonarow GC, Hammill BG, Al-Khatib SM, Yancy CW, O'Connor CM, Schulman KA, Peterson ED, Curtis LH. Clinical effectiveness of implantable cardioverter-defibrillators among medicare beneficiaries with heart failure. Circ Heart Fail. 2010 Jan;3(1):7-13. doi: 10.1161/CIRCHEARTFAILURE.109.884395. Epub 2009 Dec 15. PMID 20009044
- [Derived] Fonarow GC, Abraham WT, Albert NM, Stough WG, Gheorghiade M, Greenberg BH, O'Connor CM, Nunez E, Yancy CW, Young JB. Day of admission and clinical outcomes for patients hospitalized for heart failure: findings from the Organized Program to Initiate Lifesaving Treatment in Hospitalized Patients With Heart Failure (OPTIMIZE-HF). Circ Heart Fail. 2008 May;1(1):50-7. doi: 10.1161/CIRCHEARTFAILURE.107.748376. PMID 19808270
- [Derived] Fonarow GC, Abraham WT, Albert NM, Stough WG, Gheorghiade M, Greenberg BH, O'Connor CM, Sun JL, Yancy C, Young JB; OPTIMIZE-HF Investigators and Hospitals. Age- and gender-related differences in quality of care and outcomes of patients hospitalized with heart failure (from OPTIMIZE-HF). Am J Cardiol. 2009 Jul 1;104(1):107-15. doi: 10.1016/j.amjcard.2009.02.057. PMID 19576329
- [Derived] Flaherty JD, Rossi JS, Fonarow GC, Nunez E, Stough WG, Abraham WT, Albert NM, Greenberg BH, O'Connor CM, Yancy CW, Young JB, Davidson CJ, Gheorghiade M. Influence of coronary angiography on the utilization of therapies in patients with acute heart failure syndromes: findings from Organized Program to Initiate Lifesaving Treatment in Hospitalized Patients with Heart Failure (OPTIMIZE-HF). Am Heart J. 2009 Jun;157(6):1018-25. doi: 10.1016/j.ahj.2009.03.011. Epub 2009 Apr 23. PMID 19464412
- [Derived] Hammill BG, Hernandez AF, Peterson ED, Fonarow GC, Schulman KA, Curtis LH. Linking inpatient clinical registry data to Medicare claims data using indirect identifiers. Am Heart J. 2009 Jun;157(6):995-1000. doi: 10.1016/j.ahj.2009.04.002. PMID 19464409
- [Derived] O'Connor CM, Abraham WT, Albert NM, Clare R, Gattis Stough W, Gheorghiade M, Greenberg BH, Yancy CW, Young JB, Fonarow GC. Predictors of mortality after discharge in patients hospitalized with heart failure: an analysis from the Organized Program to Initiate Lifesaving Treatment in Hospitalized Patients with Heart Failure (OPTIMIZE-HF). Am Heart J. 2008 Oct;156(4):662-73. doi: 10.1016/j.ahj.2008.04.030. PMID 18926148
- [Derived] Abraham WT, Fonarow GC, Albert NM, Stough WG, Gheorghiade M, Greenberg BH, O'Connor CM, Sun JL, Yancy CW, Young JB; OPTIMIZE-HF Investigators and Coordinators. Predictors of in-hospital mortality in patients hospitalized for heart failure: insights from the Organized Program to Initiate Lifesaving Treatment in Hospitalized Patients with Heart Failure (OPTIMIZE-HF). J Am Coll Cardiol. 2008 Jul 29;52(5):347-56. doi: 10.1016/j.jacc.2008.04.028. PMID 18652942
- [Derived] Fonarow GC, Abraham WT, Albert NM, Stough WG, Gheorghiade M, Greenberg BH, O'Connor CM, Sun JL, Yancy CW, Young JB; OPTIMIZE-HF Investigators and Coordinators. Influence of beta-blocker continuation or withdrawal on outcomes in patients hospitalized with heart failure: findings from the OPTIMIZE-HF program. J Am Coll Cardiol. 2008 Jul 15;52(3):190-9. doi: 10.1016/j.jacc.2008.03.048. PMID 18617067
- [Derived] Fonarow GC, Abraham WT, Albert NM, Stough WG, Gheorghiade M, Greenberg BH, O'Connor CM, Nunez E, Yancy CW, Young JB. A smoker's paradox in patients hospitalized for heart failure: findings from OPTIMIZE-HF. Eur Heart J. 2008 Aug;29(16):1983-91. doi: 10.1093/eurheartj/ehn210. Epub 2008 May 15. PMID 18487210
- [Derived] Fonarow GC, Abraham WT, Albert NM, Stough WG, Gheorghiade M, Greenberg BH, O'Connor CM, Pieper K, Sun JL, Yancy CW, Young JB; OPTIMIZE-HF Investigators and Hospitals. Factors identified as precipitating hospital admissions for heart failure and clinical outcomes: findings from OPTIMIZE-HF. Arch Intern Med. 2008 Apr 28;168(8):847-54. doi: 10.1001/archinte.168.8.847. PMID 18443260
- [Derived] Yancy CW, Abraham WT, Albert NM, Clare R, Stough WG, Gheorghiade M, Greenberg BH, O'Connor CM, She L, Sun JL, Young JB, Fonarow GC. Quality of care of and outcomes for African Americans hospitalized with heart failure: findings from the OPTIMIZE-HF (Organized Program to Initiate Lifesaving Treatment in Hospitalized Patients With Heart Failure) registry. J Am Coll Cardiol. 2008 Apr 29;51(17):1675-84. doi: 10.1016/j.jacc.2008.01.028. PMID 18436120
- [Derived] Young JB, Abraham WT, Albert NM, Gattis Stough W, Gheorghiade M, Greenberg BH, O'Connor CM, She L, Sun JL, Yancy CW, Fonarow GC; OPTIMIZE-HF Investigators and Coordinators. Relation of low hemoglobin and anemia to morbidity and mortality in patients hospitalized with heart failure (insight from the OPTIMIZE-HF registry). Am J Cardiol. 2008 Jan 15;101(2):223-30. doi: 10.1016/j.amjcard.2007.07.067. PMID 18178411
- [Derived] Fonarow GC, Abraham WT, Albert NM, Stough WG, Gheorghiade M, Greenberg BH, O'Connor CM, Sun JL, Yancy CW, Young JB; OPTIMIZE-HF Investigators and Coordinators. Prospective evaluation of beta-blocker use at the time of hospital discharge as a heart failure performance measure: results from OPTIMIZE-HF. J Card Fail. 2007 Nov;13(9):722-31. doi: 10.1016/j.cardfail.2007.06.727. PMID 17996820
- [Derived] Fonarow GC, Stough WG, Abraham WT, Albert NM, Gheorghiade M, Greenberg BH, O'Connor CM, Sun JL, Yancy CW, Young JB; OPTIMIZE-HF Investigators and Hospitals. Characteristics, treatments, and outcomes of patients with preserved systolic function hospitalized for heart failure: a report from the OPTIMIZE-HF Registry. J Am Coll Cardiol. 2007 Aug 21;50(8):768-77. doi: 10.1016/j.jacc.2007.04.064. Epub 2007 Aug 6. PMID 17707182
- [Derived] Fonarow GC, Abraham WT, Albert NM, Gattis Stough W, Gheorghiade M, Greenberg BH, O'Connor CM, Pieper K, Sun JL, Yancy CW, Young JB; OPTIMIZE-HF Investigators and Hospitals. Influence of a performance-improvement initiative on quality of care for patients hospitalized with heart failure: results of the Organized Program to Initiate Lifesaving Treatment in Hospitalized Patients With Heart Failure (OPTIMIZE-HF). Arch Intern Med. 2007 Jul 23;167(14):1493-502. doi: 10.1001/archinte.167.14.1493. PMID 17646603
- [Derived] Greenberg BH, Abraham WT, Albert NM, Chiswell K, Clare R, Stough WG, Gheorghiade M, O'Connor CM, Sun JL, Yancy CW, Young JB, Fonarow GC. Influence of diabetes on characteristics and outcomes in patients hospitalized with heart failure: a report from the Organized Program to Initiate Lifesaving Treatment in Hospitalized Patients with Heart Failure (OPTIMIZE-HF). Am Heart J. 2007 Aug;154(2):277.e1-8. doi: 10.1016/j.ahj.2007.05.001. PMID 17643576
- [Derived] Albert NM, Fonarow GC, Abraham WT, Chiswell K, Stough WG, Gheorghiade M, Greenberg BH, O'Connor CM, Sun JL, Yancy CW, Young JB. Predictors of delivery of hospital-based heart failure patient education: a report from OPTIMIZE-HF. J Card Fail. 2007 Apr;13(3):189-98. doi: 10.1016/j.cardfail.2006.11.008. PMID 17448416
- [Derived] Fonarow GC, Abraham WT, Albert NM, Stough WG, Gheorghiade M, Greenberg BH, O'Connor CM, Sun JL, Yancy C, Young JB; OPTIMIZE-HF Investigators and Coordinators. Carvedilol use at discharge in patients hospitalized for heart failure is associated with improved survival: an analysis from Organized Program to Initiate Lifesaving Treatment in Hospitalized Patients with Heart Failure (OPTIMIZE-HF). Am Heart J. 2007 Jan;153(1):82.e1-11. doi: 10.1016/j.ahj.2006.10.008. PMID 17174643